CLINICAL TRIAL: NCT06601036
Title: Sevoflurane Sedation as an Alternative for Awake Fiberoptic Intubation in Difficult Airway Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Marwa Ahmed Abogabal, Lecturer of Anesthesiology, Intensive Care and Pain, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR591/3/24
Record Dates: First submitted 2024-09-14; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Sevoflurane; Sedation; Awake Fiberoptic Intubation; Difficult Airway
MeSH Terms: interventions — Sevoflurane; Lidocaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane sedation group (Experimental): Patients will undergo fiberoptic intubation under sevoflurane sedation.
  Interventions: Drug: Sevoflurane
- Awake fiberoptic group (Active Comparator): Patients will undergo fiberoptic intubation with bilateral Superior Laryngeal Nerve block and Recurrent laryngeal nerve block.
  Interventions: Drug: 2% Xylocaine (2 ml )

INTERVENTIONS:
Drug: Sevoflurane — Patients will undergo fiberoptic intubation under sevoflurane sedation.
  Arms: Sevoflurane sedation group
Drug: 2% Xylocaine (2 ml ) — Patients will undergo fiberoptic intubation with bilateral Superior Laryngeal Nerve block and Recurrent laryngeal nerve block.
  Arms: Awake fiberoptic group

SUMMARY:
The aim of this study is to compare patient satisfaction and intubating conditions with fiber optic intubation under sevoflurane sedation versus airway blocks in difficult airway patients

DETAILED DESCRIPTION:
Awake fiberoptic intubation (AFOI) is a suitable option for anticipated difficult intubation. The ideal condition for AFOI requires a calm, cooperative patient with blunted airway reflexes to facilitate easy intubation, especially if there is difficulty with laryngeal anatomy and/or pathology.

For this purpose, sedative and anxiolytic agents such as benzodiazepines, sevoflurane, remifentanil, ketamine, propofol, and dexmedetomidine are almost always required to relieve the patients from comfort without impairing ventilation. Patient responsiveness and cooperation are almost always required.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 50 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-II.
* Patients with difficult airway (Mallampati grade 3 and 4 with mouth opening less than 5 cm).

Exclusion Criteria:

* Patient refusal.
* Patients with bleeding disorders and nasal mass.
* Allergy or intolerance to one of the study medications.
* Patients with uncontrolled systemic diseases.
* patients with gastro-esophageal reflex.
* history of nasopharyngeal surgery or drug abuse.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Degree of patient satisfaction | Immediately after intubation
  The degree of patient satisfaction will be assessed on a 4-point Likert scale patient satisfaction (1, very dissatisfied; 2, unsatisfied; 3, satisfied; 4, very satisfied).

SECONDARY OUTCOMES:
Intubation time | Intraoperatively
  Intubation time (time from insertion of the fiberoptic bronchoscope throughout the nose till confirmation of intubation with capnography)
Heart rate | 5 minutes after intubation
  Heart rate will be recorded on arrival to the operating room as a baseline, immediately prior to fiberoptic intubation, at the time of intubation and then at 1, 3, and 5 minutes after intubation.
Mean arterial pressure | 5 minutes after intubation
  Mean arterial pressure will be recorded on arrival to the operating room as a baseline, immediately prior to fiberoptic intubation, at the time of intubation and then at 1, 3, and 5 minutes after intubation.
Patient's tolerance to endoscopy | Intraoperatively
  The patient's reaction to the placement of the fiberoptic scope will be assessed on a scale of 1 to 5 and will be recorded (1, no reaction; 2, slight grimacing; 3, severe grimacing; 4, verbal objection; 5, defensive movement of head, hands, or feet).
Patient's tolerance to intubation | Intraoperatively
  The patient's reaction to the placement of the endotracheal tube will be assessed on a scale of 1 to 5 and was recorded (1, no reaction; 2, slight grimacing; 3, severe grimacing; 4, verbal objection; 5, defensive movement of head, hands, or feet)

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.